CLINICAL TRIAL: NCT05297929
Title: Bioequivalence of Irbesartan Tablets (0.15g/Tablet) in a Randomized, Open, Two-cycle, Two-crossover Single Fasting/Postprandial State in Healthy Subjects
Brief Title: A Bioequivalence Trial of Irbesartan Tablets（0.15g） in Healthy Chinese Subjects
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Affiliated Hospital of Qingdao University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: BJK-BE-EBST-2021017-ZJHH
Record Dates: First submitted 2022-03-06; First posted 2022-03-28 (Actual); Last update posted 2022-03-28 (Actual); Status verified 2022-03

CONDITIONS: Irbesartan Tablets (0.15g/Tablet); Under Fasted Condition; Under Fed Condition; Bioequivalence
MeSH Terms: interventions — Irbesartan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: Reference formulation (Experimental): Irbesartan tablet (0.15g/tablet) , Manufacturer: Sanofi Winthrop Industries
  Interventions: Drug: Irbesartan Tablet
- Experimental: Test formulation (Experimental): Irbesartan tablet (0.15g/tablet) , Manufacturer: Zhejiang Hua Hai Pharmaceutical Co. LTD
  Interventions: Drug: Irbesartan Tablet

INTERVENTIONS:
Drug: Irbesartan Tablet — Drug: Irbesartan Oral administration on an empty stomach／fed condition

SUMMARY:
To study the pharmacokinetics of test preparation and reference preparation irbesartan tablets (0.15g/tablet) in a single oral administration in fasting and fed state,respectively, in healthy adult subjects, and to evaluate the bioequivalence of the two preparations

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male and female subjects aged 18 to 45 years (inclusive);
2. Male subjects not less than 50 kg weight, women were not less than 45 kg weight. Scope of body mass index (BMI) of 19.0 ~ 26.0 kg/m2 / BMI = weight (kg)/height (m) 2] (including 19.0 and 26.0);
3. Have the ability to communicate with normal researchers/staff and comply with the relevant provisions on the administration of hospital;
4. The subject fully understands the purpose, nature, methods and possible adverse reactions of the test, voluntarily acts as a subject, and signs an informed consent before the start of any study program;
5. Participants must agree on the non-drug contraception and begin screening and the last time the medicine to prevent pregnancy or within 6 months after with couple of pregnancy.

Exclusion Criteria:

1. The respiratory system, circulatory system, digestive system, urinary system, blood system, endocrine system, immune system, nervous system, spirit, system and metabolic abnormalities any clinical history of serious illness, or any other disease which can interfere with the test results or physiological conditions and the researchers judged as abnormal have clinical significance;
2. The physical examination, vital signs, abnormal electrocardiogram (ecg) and laboratory examination (unless approved by the researchers determine abnormal no clinical significance).
3. Have difficulty swallowing or any affect drug absorption of gastrointestinal diseases history or has a history of digestive surgery, hemorrhoids surgery (appendix except and abdomen ditch hernia repair surgery) or affect the pharmacokinetic factors are known;
4. A history of orthostatic hypotension or screening phase orthostatic hypotension;
5. In the past year of alcohol abuse, such as drinking more than 14 units of alcohol a week (1 unit of alcohol is equal to 360 ml 150 ml beer or wine or 45 ml 40% distillation wine, such as the spirit Erguotou, etc.) or the whole experiments cannot stop drinkers;
6. 3 months prior to screening the average daily amount of more than 5 pieces, or cannot be confirmed and agreed to the first cycle dosing 48 hours before the last time to collect blood before smoking;
7. Human immunodeficiency virus (HIV), hepatitis b surface antigen, treponema pallidum antibody or hepatitis c virus (HCV) antibody is positive;
8. Alcohol breath test or drug abuse inspection is positive;
9. The first cycle within 3 months before the treatment, attend a group into any clinical trials;
10. Within a month before the first cycle to use any other drugs, including prescription drugs or over-the-counter medications (including oral multivitamins, herb medicine, Chinese medicine, medicine stewed food or dietary supplements);
11. Subjects were unable to confirm and agree with the first cycle 48 hours before delivery to the front of the last blood ban suits oranges, grapefruits, grapefruit, pomelo, orange, or any alcoholic, xanthine and caffeine foods and beverages, including chocolate, tea, coffee, coke, etc.);
12. This product and its analogues, or to any known a complementary makings allergy, or appeared to two or more drugs, such as food allergies or allergic constitution;
13. There are galactose intolerance, total lactase deficiency or glucose - galactose malabsorption of rare genetic disease;
14. Cannot accept venous blood collection or meals provided by the clinical trial center;
15. Drug delivery within one month before the first cycle vaccinated;
16. The first cycle for three months before donating blood or blood loss is equal to or more than 400 mL;
17. Pregnant or breastfeeding women, or screening in the first two weeks of women with and without protective behavior;
18. The researchers determine the subjects are not suitable for participating in this study or for other reasons can not complete the study subjects

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 54 (Estimated)
Dates: Start 2022-02-17 (Actual); Primary Completion 2022-04-09 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
AUC0-t | up to 1 year
  Pharmacokinetic parameter AUC0-t estimated by non-compartmental analysis model based on the plasma concentration data of concentration data of irbesartan
AUC0-∞ | up to 1 year
  Pharmacokinetic parameter AUC0-∞ estimated by non-compartmental analysis model based on the plasma concentration data of concentration data of irbesartan
Cmax | up to 1 year
  Pharmacokinetic parameter Cmax estimated by non-compartmental analysis model based on the plasma concentration data of concentration data of irbesartan
Tmax | up to 1 year
  Pharmacokinetic parameter Tmax estimated by non-compartmental analysis model based on the plasma concentration data of concentration data of irbesartan
bioequivalence | up to 1 year
  Analysis of variance (ANOVA) was performed after logarithmic conversion of main pharmacokinetic parameters (Cmax, AUC) to calculate 90% confidence interval of geometric mean ratio of main pharmacokinetic parameters of the two preparations, and equivalence comparison was conducted. The equivalent interval was set to 80.00%~125.00%

SECONDARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE | up to 6 months
  Number of participants with treatment-related adverse events as assessed by CTCAE

CONTACTS AND LOCATIONS:
Overall Officials: Yu Cao, professor, Principal Investigator — The Affiliated Hospital of Qingdao University
Locations (1):
- The Affiliated Hospital of Qingdao University, Qingdao, Shandong, China

IPD SHARING:
Plan to Share IPD: No